CLINICAL TRIAL: NCT05584917
Title: Physical Activity Return After Popliteal Artery Entrapement Syndrome Surgery With Tegner Activity Scale
Brief Title: Physical Activity Return After Popliteal Artery Entrapement Syndrome Surgery
Acronym: PAES
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 49RC22_0305
Record Dates: First submitted 2022-10-11; First posted 2022-10-18 (Actual); Last update posted 2022-12-29 (Actual); Status verified 2022-10

CONDITIONS: Popliteal Artery Entrapment
MeSH Terms: conditions — Popliteal Artery Entrapment Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- surgery patient (Experimental): phone call after surgery to answer the tegner activity scale
  Interventions: Behavioral: tegner acticity scale

INTERVENTIONS:
Behavioral: tegner acticity scale — phone call to complete the tegner activity scale after surgery

SUMMARY:
evaluation of physical activity return after popliteal artery entrapement syndrome surgery with the tegner activity scale

ELIGIBILITY:
Inclusion Criteria:

* popliteal artery entrapement syndrome surgery between 2010 and 2020 at the university center of Angers

Exclusion Criteria:

* denied to participate

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-06-11 (Estimated); Study Completion 2024-02-28 (Estimated)

PRIMARY OUTCOMES:
comparison | change from baseline of the tegner activity scale 1 year after surgery
  comparison between tegner activity scale results before and after surgery. Tegner activity scale is from 0 to 10, minimum 0 and maximum 10. Higher score means a better outcome

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital, Angers, France

IPD SHARING:
Plan to Share IPD: No